CLINICAL TRIAL: NCT00590122
Title: Comparison of Orally Dissolving Carbidopa/Levodopa (Parcopa) to Conventional Oral Carbidopa/Levodopa: A Single-Dose, Double-Blind, Double-Dummy, Placebo-Controlled, Crossover Trial
Brief Title: Parcopa Versus Carbidopa-levodopa in a Single Dose Cross-over Comparison Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Joseph Jankovic, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-19596
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; time to "on"; delayed on
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomization Group b (Experimental): Parcopa at equivalent dosage to subjects current stable dose
  Interventions: Drug: Parcopa
- Randomization Group a (Active Comparator): Carbidopa-levodopa (Sinemet)at subjects current stable dose
  Interventions: Drug: carbidopa-levodopa (Sinemet)

INTERVENTIONS:
Drug: Parcopa — at subjects current stable dose of comparator
  Arms: Randomization Group b
Drug: carbidopa-levodopa (Sinemet) — at subjects current stable dose
  Arms: Randomization Group a

SUMMARY:
To find out if a single dose of Parcopa®, a form of levodopa that dissolves in your mouth, works faster than regular oral levodopa which is swallowed, in fluctuating PD patients.

DETAILED DESCRIPTION:
This is a study to compare orally dissolving levodopa (Parcopa) to the conventional immediate release oral levodopa. This is a single-dose, double-blind, placebo controlled crossover trial in participants with Parkinson disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 31 and 80 -Diagnosis of idiopathic Parkinson's disease for at least three years duration
* Patients requiring levodopa for their PD
* Good subjective response to levodopa
* Fluctuating symptoms defined by wearing off phenomenon, any dyskinesia, and/or dose failures
* A UPDRS -off- motor score of at least 25
* Subjects willing to give informed consent
* Subjects who are able and willing to comply with study procedures
* If female of child-bearing potential, will use one of the approved birth control measures:

  1. Hormonal contraceptives
  2. Spermicidal and barrier
  3. Intrauterine device
  4. Partner sterility

Exclusion Criteria:

* Subjects with evidence of significant dementia
* Subjects with significant oral lesions
* History of unstable cardiac disease including angina or congestive heart failure within 3 months prior to study entry
* History of clinically significant renal disease including renal insufficiency of sufficient degree to require adjunctive treatment or dietary restrictions
* History of clinically significant hepatic disease, including previously documented cirrhosis or hepatic insufficiency or jaundice within 3 months prior to study entry.
* Subjects with poor response to levodopa
* Women who are pregnant, breast-feeding, or planning to become pregnant during this study are excluded from participation due to unknown effects of the study drug on the fetus.

Ages: 31 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Ondo, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- PDCMDC 6550 Fannin, Suite 1801, Houston, Texas, United States

REFERENCES:
- [Background] Ondo WG, Shinawi L, Moore S. Comparison of orally dissolving carbidopa/levodopa (Parcopa) to conventional oral carbidopa/levodopa: A single-dose, double-blind, double-dummy, placebo-controlled, crossover trial. Mov Disord. 2010 Dec 15;25(16):2724-7. doi: 10.1002/mds.23158. PMID 20925074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Crossover study design
Groups:
- B-Parcopa Arm First Then Crossover to Carbidopa/Levodopa Arm: Parcopa: at subjects current stable dose of comparator first (Day 1) then crossover to the carbidopa/levodopa arm (Day 2)
- A-Carbidopa/Levodopa Arm Then Crossover to Parcopa Arm: carbidopa-levodopa at subjects current stable dose (Day 1) then crossover to the parcopa comparator arm of the study (Day 2)
Period: Overall Study
Arm/Group | B-Parcopa Arm First Then Crossover to Carbidopa/Levodopa Arm | A-Carbidopa/Levodopa Arm Then Crossover to Parcopa Arm
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — swallowed oral dissolving dose | 1 | 0

BASELINE CHARACTERISTICS:
Population: Crossover design study total number same in each group
Groups:
- B-Parcopa Arm First Then Crossover to Carbidopa/Levodopa Arm: Parcopa: at subjects current stable dose of comparator
- A-Carbidopa/Levodopa Arm Then Crossover to Parcopa Arm: carbidopa-levodopa at subjects current stable dose
- Total: Total of all reporting groups
Arm/Group | B-Parcopa Arm First Then Crossover to Carbidopa/Levodopa Arm | A-Carbidopa/Levodopa Arm Then Crossover to Parcopa Arm | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 7 | 8 | 15
  Hispanic | 2 | 1 | 3
  African-American | 1 | 0 | 1
  Asian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Time in Minutes From When a Patient Was in a Clinical "Off" State, Took Their Medication and Went Into a Clinical "on" State
Description: Time to "on" state (benefit with regard to mobility, stiffness and slowness) with parcopa versus carbidopa/levodopa immediate release compound. This measurement is compared between Parcopa and carbidopa/levodopa wit the first morning dose of each intervention. Study duration was 2 days.
Time Frame: first dose of day for each arm
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- B-Parcopa Arm: Parcopa: at subjects current stable dose of comparator
- A-Carbidopa/Levodopa Arm: carbidopa-levodopa at subjects current stable dose
Arm/Group | B-Parcopa Arm | A-Carbidopa/Levodopa Arm
Number analyzed (Participants) | 20 | 20
minutes | 23.9 (9.9) | 28.5 (19.4)

ADVERSE EVENTS:
Time Frame: 2 day, double blind crossover study
Arm/Group | B-Parcopa Arm | A-Carbidopa/Levodopa Arm
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-Parcopa Arm (N=20) | A-Carbidopa/Levodopa Arm (N=20)
dyskinesia (General disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No